CLINICAL TRIAL: NCT05512663
Title: A Pilot Study Evaluating Safety and Efficacy of Transperineal Focal Irreversible Electroporation (IRE) of Anterior Prostate Cancer in Patients With an Intermediate Risk.
Brief Title: Safety and Efficacy Evaluation of Transperineal Irreversible Electroporation (IRE) of Anterior Prostate Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Maurice Anidjar,MD, Associate Professor, Division of Urology,MD,PhD, Jewish General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-2815
Record Dates: First submitted 2021-04-06; First posted 2022-08-23 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Prostate Cancer
Keywords: Intermediate Risk Prostate Cancer; Irreversible Electroporation (IRE)
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Electroporation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Irreversible Electroporation (IRE) treatment (Experimental): Focal Irreversible Electroporation (IRE) delivered by NanoKnife System is composed of the NanoKnife Generator and NanoKnife Single Electrode Probes.With the NanoKnife System, electrical current is delivered between pairs of probes in a series of pulses. The waveform of the current is adjustable as determined by clinician chosen parameters. Up to six probes may be placed in an array within the tissue. The probes of the array are matched as pairs by the system. When probes are activated via a foot pedal, the scheduled current is delivered to tissue between subsequent pairs of probes. Soft tissue between the probes is ablated.
  Interventions: Device: Irreversible Electroporation (IRE)

INTERVENTIONS:
Device: Irreversible Electroporation (IRE) — The area of the prostate that was positive for cancer based on the transperineal prostate biopsy will be targeted for ablation via the NanoKnife System. An MRI/TRUS fusion device probe will be placed in the rectum and the prostate will be visualized in both sagittal and axial views. The ultrasound grid which was used during the mapping biopsy will be oriented using anatomical landmarks and used to identify the location of the positive biopsy cores. The NanoKnife Single Electrode Probes will be surgically inserted into the prostate through the perineum using MRI/TRUS fusion guidance and the ultrasound grid for guidance.

SUMMARY:
Most prostate cancer treatment research in the last decade has been focused on trying to improve quality of life, while maintaining a high level of cancer control. However, the concept of Focal treatment is proposed as an intermediate option between active surveillance and treatment of the whole prostate. Focal ablation aims to efficiently treat the localized cancer while reducing complications related to standard treatments, including the risks of incontinence and impotence.

Focal Irreversible Electroporation (IRE) delivered by NanoKnife System is composed of the NanoKnife Generator and NanoKnife Single Electrode Probes. With IRE, an electrical current is delivered between a pair of probes in a series of pulses. These pulses create irreversible pores in cell membranes and lead to cell death which allow for only the tissue between these probes being destroyed.

The aim of this study is to analyze the safety and efficacy of transperineal IRE treatments in intermediate risk anteriorly localized prostate cancer patients.

DETAILED DESCRIPTION:
There are different effective treatment options for intermediate risk prostate cancer to choose from. The standard of care are definite treatments such as robotic surgery or radiotherapy. Robotic surgeries involve the removal of the entire prostate. On the other hand, radiotherapy is a form of treatment that is done by either an external beam at high and low dose rate or by brachytherapy. The external beam at high or low dose rate targets the entire prostate. Brachytherapy, which involves a special radiation source that is placed inside the tumour, targets only specific parts of the prostate.

Both robotic surgeries and radiotherapy provide a greater certainty of cancer control than any other treatments option, however there is a significant risk of side effects that many follow these treatments. Among which, there is a 50% likelihood for impotence, 5-10% likelihood of incontinence and 5-20% likelihood of bowel dysfunction.

One way of reducing the unwanted side-effects from radical treatment of prostate cancer may be to direct treatment to only areas of the cancer. This is called focal therapy, which is the form of treatment that will be performed and observed in this study. There has been recent research done on focal therapies that have been shown to be more advantageous than having radical therapy or radiotherapy. Some of these advantages include: decrease of chance or elimination of possible side-effects post-treatment, it is a less invasive treatment option and the omission of overnight hospital stay post-treatment, among others.

This study is designed to look at an experimental treatment of localized prostate cancer by Focal Irreversible Electroporation (IRE) delivered by the NanoKnife System.

ELIGIBILITY:
Inclusion Criteria:

* 1. Has at least a 10 year life expectancy 2. Have histologically confirmed organ-confined prostate cancer - clinical Stage T1-T2c N0M0 3. Have a PSA <=15ng/mL 4. Has Gleason <=7 (4+3 or 3+4) 5. Has maximum cancer core length >=4mm 6. No evidence of extraprostatic extension or seminal vesicle invasion by mpMRI 7. Able to visualize prostate gland adequately on transrectal ultrasound imaging during enrollment evaluation 8. Transperineal prostate biopsies (template mapping and/or limited targeted) correlating with clinically significant lesion in the area of the MR-visible lesion (within 2 Barzell zones) 9. A visible lesion on mpMRI, that is accessible to IRE treatment 10. Must sign a written informed consent 11. Understands and accepts the obligation and is logistically able to present for all scheduled follow-up visits

Exclusion Criteria:

* 1. Have known hypersensitivity to pancuronium bromide, atricurium or cisatricurium 2. Unfit for anthesthia or have a contraindication for agents listed for paralysis 3. Have an active urinary tract infection (UTI) 4. Have a history of bladder neck contracture 5. Are interested in future fertility 6. Have a history (within 3 years) of inflammatory bowel disease 7. Have a concurrent major debilitating illness 8. Had a malignancy, other than prostate or skin cancer (except malignant melanoma), within 5 years 9. Have any active implanted electronic device (eg, pacemaker) 10. Are unable to catheterize due to a urethral stricture disease 11. Have had prior or current prostate cancer therapies:

  1. Biologic therapy for prostate cancer
  2. Chemotherapy for prostate cancer
  3. Hormonal therapy for prostate cancer within three months of procedure
  4. Radiotherapy for prostate cancer
  5. Surgery for prostate cancer 12. Have had prior transurethral prostatectomy (TURP), or urethral stent 13. Have had prior major rectal surgery (except hemorrhoids) 14. Unfit for pelvic MRI scanning (e.g. severe claustrophobia, permanent cardiac pacemaker, metallic implant etc… likely to contribute significant artefact to images) 15. Have a non-visible tumor on mpMRI

Ages: 18 Years to 95 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
The occurrence of possible Adverse Events | From the operation date until the end of the study (12 months)
  The complete description of any possible Adverse Events or Serious Adverse Events, including: Incidence, Type, Duration, Severity and Relationship to the study device.
Analysis of Urinary function by UCLA-EPIC scores #1.1 | At Screening (Pre-operative)
  The University of California, Los Angeles - Expanded Prostate Cancer Index Composite score will be evaluated. UCLA-EPIC is a 26-question short form as a Standard Set of patient-centered outcome for men with both localized and advanced prostate cancer. The 5 domains of questions: Urinary Incontinence, Urinary Irritative/Obstructive, Bowel, Sexual, and Hormonal.
  Response options for each EPIC item form a Likert scale, and multi-item scale scores are transformed linearly to a 0-100 scale with higher scores representing better Health Related Quality of Life (HRQOL).
Analysis of Urinary function by UCLA-EPIC scores #1.2 | At 1-month post-operation
  The University of California, Los Angeles - Expanded Prostate Cancer Index Composite score will be evaluated. UCLA-EPIC is a 26-question short form as a Standard Set of patient-centered outcome for men with both localized and advanced prostate cancer. The 5 domains of questions: Urinary Incontinence, Urinary Irritative/Obstructive, Bowel, Sexual, and Hormonal.
  Response options for each EPIC item form a Likert scale, and multi-item scale scores are transformed linearly to a 0-100 scale with higher scores representing better Health Related Quality of Life (HRQOL).
Analysis of Urinary function by UCLA-EPIC scores #1.3 | At 3-month post-operation
  The University of California, Los Angeles - Expanded Prostate Cancer Index Composite score will be evaluated. UCLA-EPIC is a 26-question short form as a Standard Set of patient-centered outcome for men with both localized and advanced prostate cancer. The 5 domains of questions: Urinary Incontinence, Urinary Irritative/Obstructive, Bowel, Sexual, and Hormonal.
  Response options for each EPIC item form a Likert scale, and multi-item scale scores are transformed linearly to a 0-100 scale with higher scores representing better Health Related Quality of Life (HRQOL).
Analysis of Urinary function by UCLA-EPIC scores #1.4 | At 6-month post-operation
  The University of California, Los Angeles - Expanded Prostate Cancer Index Composite score will be evaluated. UCLA-EPIC is a 26-question short form as a Standard Set of patient-centered outcome for men with both localized and advanced prostate cancer. The 5 domains of questions: Urinary Incontinence, Urinary Irritative/Obstructive, Bowel, Sexual, and Hormonal.
  Response options for each EPIC item form a Likert scale, and multi-item scale scores are transformed linearly to a 0-100 scale with higher scores representing better Health Related Quality of Life (HRQOL).
Analysis of Urinary function by UCLA-EPIC scores #1.5 | At 9-month post-operation
  The University of California, Los Angeles - Expanded Prostate Cancer Index Composite score will be evaluated. UCLA-EPIC is a 26-question short form as a Standard Set of patient-centered outcome for men with both localized and advanced prostate cancer. The 5 domains of questions: Urinary Incontinence, Urinary Irritative/Obstructive, Bowel, Sexual, and Hormonal.
  Response options for each EPIC item form a Likert scale, and multi-item scale scores are transformed linearly to a 0-100 scale with higher scores representing better Health Related Quality of Life (HRQOL).
Analysis of Urinary function by UCLA-EPIC scores #1.6 | At 12-month post-operation
  The University of California, Los Angeles - Expanded Prostate Cancer Index Composite score will be evaluated. UCLA-EPIC is a 26-question short form as a Standard Set of patient-centered outcome for men with both localized and advanced prostate cancer. The 5 domains of questions: Urinary Incontinence, Urinary Irritative/Obstructive, Bowel, Sexual, and Hormonal.
  Response options for each EPIC item form a Likert scale, and multi-item scale scores are transformed linearly to a 0-100 scale with higher scores representing better Health Related Quality of Life (HRQOL).
Analysis of Urinary function by IPSS-QoL scores #2.1 | At Screening (Pre-operative)
  The International Prostate Symptom Score-Quality of Life (IPSS-QoL) score will be evaluated. The IPSS-QoL is based on the answers to seven questions concerning urinary symptoms and one question concerning quality of life. The answers are assigned points from 0 to 5. The total score can therefore range from 0 to 35 (asymptomatic to very symptomatic).
  The American Urological Association (AUA) Symptom Index which currently categorizes symptoms as follows:
  Mild (symptom score less than of equal to 7) Moderate (symptom score range 8-19) Severe (symptom score range 20-35)
  A low score will produce better outcomes.
Analysis of Urinary function by IPSS-QoL scores #2.2 | At 1-month post-operation
  The International Prostate Symptom Score-Quality of Life (IPSS-QoL) score will be evaluated. The IPSS-QoL is based on the answers to seven questions concerning urinary symptoms and one question concerning quality of life. The answers are assigned points from 0 to 5. The total score can therefore range from 0 to 35 (asymptomatic to very symptomatic).
  The American Urological Association (AUA) Symptom Index which currently categorizes symptoms as follows:
  Mild (symptom score less than of equal to 7) Moderate (symptom score range 8-19) Severe (symptom score range 20-35)
  A low score will produce better outcomes.
Analysis of Urinary function by IPSS-QoL scores #2.3 | At 3-month post-operation
  The International Prostate Symptom Score-Quality of Life (IPSS-QoL) score will be evaluated. The IPSS-QoL is based on the answers to seven questions concerning urinary symptoms and one question concerning quality of life. The answers are assigned points from 0 to 5. The total score can therefore range from 0 to 35 (asymptomatic to very symptomatic).
  The American Urological Association (AUA) Symptom Index which currently categorizes symptoms as follows:
  Mild (symptom score less than of equal to 7) Moderate (symptom score range 8-19) Severe (symptom score range 20-35)
  A low score will produce better outcomes.
Analysis of Urinary function by IPSS-QoL scores #2.4 | At 6-month post-operation
  The International Prostate Symptom Score-Quality of Life (IPSS-QoL) score will be evaluated. The IPSS-QoL is based on the answers to seven questions concerning urinary symptoms and one question concerning quality of life. The answers are assigned points from 0 to 5. The total score can therefore range from 0 to 35 (asymptomatic to very symptomatic).
  The American Urological Association (AUA) Symptom Index which currently categorizes symptoms as follows:
  Mild (symptom score less than of equal to 7) Moderate (symptom score range 8-19) Severe (symptom score range 20-35)
  A low score will produce better outcomes.
Analysis of Urinary function by IPSS-QoL scores #2.5 | At 9-month post-operation
  The International Prostate Symptom Score-Quality of Life (IPSS-QoL) score will be evaluated. The IPSS-QoL is based on the answers to seven questions concerning urinary symptoms and one question concerning quality of life. The answers are assigned points from 0 to 5. The total score can therefore range from 0 to 35 (asymptomatic to very symptomatic).
  The American Urological Association (AUA) Symptom Index which currently categorizes symptoms as follows:
  Mild (symptom score less than of equal to 7) Moderate (symptom score range 8-19) Severe (symptom score range 20-35)
  A low score will produce better outcomes.
Analysis of Urinary function by IPSS-QoL scores #2.6 | At 12-month post-operation
  The International Prostate Symptom Score-Quality of Life (IPSS-QoL) score will be evaluated. The IPSS-QoL is based on the answers to seven questions concerning urinary symptoms and one question concerning quality of life. The answers are assigned points from 0 to 5. The total score can therefore range from 0 to 35 (asymptomatic to very symptomatic).
  The American Urological Association (AUA) Symptom Index which currently categorizes symptoms as follows:
  Mild (symptom score less than of equal to 7) Moderate (symptom score range 8-19) Severe (symptom score range 20-35)
  A low score will produce better outcomes.
Analysis of Erectile function by IIEF-15 scores #1.1 | At Screening (Pre-operative)
  The International Index of Erectile Function (IIEF-15) score will be evaluated. A score of 0-5 is awarded to each of the 15 questions that examine the 4 main domains of male sexual function: erectile function, orgasmic function, sexual desire and intercourse satisfaction.
  A higher score will produce better outcomes.
Analysis of Erectile function by IIEF-15 scores #1.2 | At 1-month post-operation
  The International Index of Erectile Function (IIEF-15) score will be evaluated. A score of 0-5 is awarded to each of the 15 questions that examine the 4 main domains of male sexual function: erectile function, orgasmic function, sexual desire and intercourse satisfaction.
  A higher score will produce better outcomes.
Analysis of Erectile function by IIEF-15 scores #1.3 | At 3-month post-operation
  The International Index of Erectile Function (IIEF-15) score will be evaluated. A score of 0-5 is awarded to each of the 15 questions that examine the 4 main domains of male sexual function: erectile function, orgasmic function, sexual desire and intercourse satisfaction.
  A higher score will produce better outcomes.
Analysis of Erectile function by IIEF-15 scores #1.4 | At 6-month post-operation
  The International Index of Erectile Function (IIEF-15) score will be evaluated. A score of 0-5 is awarded to each of the 15 questions that examine the 4 main domains of male sexual function: erectile function, orgasmic function, sexual desire and intercourse satisfaction.
  A higher score will produce better outcomes.
Analysis of Erectile function by IIEF-15 scores #1.5 | At 9-month post-operation
  The International Index of Erectile Function (IIEF-15) score will be evaluated. A score of 0-5 is awarded to each of the 15 questions that examine the 4 main domains of male sexual function: erectile function, orgasmic function, sexual desire and intercourse satisfaction.
  A higher score will produce better outcomes.
Analysis of Erectile function by IIEF-15 scores #1.6 | At 12-month post-operation
  The International Index of Erectile Function (IIEF-15) score will be evaluated. A score of 0-5 is awarded to each of the 15 questions that examine the 4 main domains of male sexual function: erectile function, orgasmic function, sexual desire and intercourse satisfaction.
  A higher score will produce better outcomes.

IPD SHARING:
Plan to Share IPD: No